CLINICAL TRIAL: NCT06617494
Title: The Role of Endogenous Pain Inhibition Deficiency in Chronic TMD Pain Pathophysiology
Brief Title: Endogenous Pain Inhibition Deficiency in Chronic TMD Pain
Acronym: TMD-CPM
Status: Recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00022663
Record Dates: First submitted 2024-09-24; First posted 2024-09-27 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Chronic Temporomandibular Disorders (TMD)
Keywords: Temporomandibular disorders (TMD); Chronic pain; Healthy volunteers
MeSH Terms: conditions — Temporomandibular Joint Disorders; Chronic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic Temporomandibular disorder (TMD) pain group
  Interventions: Other: Pain modulation testing
- Age- and sex-matched pain-free controls
  Interventions: Other: Pain modulation testing

INTERVENTIONS:
Other: Pain modulation testing — During the visit, noxious heat stimuli will be applied bilaterally to the face and distant body sites as part of conditioned pain modulation (CPM) testing. The test stimuli will be individually tailored to be moderately painful, while the conditioning stimulus will vary in intensity: moderately painful, non-painful, and sham heat. Participants will also record daily TMD pain intensity ratings for seven days before and after the visit.

SUMMARY:
Temporomandibular disorders (TMDs) involve a range of conditions with varied causes, affecting a large portion of the U.S. population and posing challenges for diagnosis and management, especially in chronic cases. Despite advances in understanding TMD pathophysiology, the role of central sensitization, particularly deficient endogenous pain inhibition, remains unclear. The conditioned pain modulation (CPM) test, used to assess pain inhibition in chronic TMD pain, has produced inconsistent results due to varying testing parameters. The proposed cross-sectional study will investigate the efficiency of endogenous pain inhibition in individuals with chronic TMD pain compared to controls by applying noxious and non-noxious stimuli to facial and non-facial sites. The findings aim to clarify the impact of weaker pain inhibition over the face, how the conditioning stimulus' painfulness affects inhibition and the relationship between pain inhibition and fluctuations in TMD pain intensity.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this study, an individual must meet all the following criteria:

1. Provide informed consent, documented in a signed and dated form.
2. Will comply with all study procedures, including daily ratings filling before and after the in-person study visit, and be available for the study duration.
3. All participants of both genders between ages 18 to 74 years.
4. Cases and controls will be matched for age within ±5 years, and all participants must understand English commands to follow study procedures (e.g., during CPM testing).

Pain-free controls:

1. Age matching (within ±5 years)
2. No previous diagnosis for the most common pain-related TMD as defined in the DC/TMD criteria (myalgia, arthralgia, headache attributed to TMD)
3. No significant orofacial pain (jaw pain, TMJ pain) in the past 3 months (""significant"" meaning 5 or more days in any month or any pain during the past month)
4. No report of significant pain in the last 3 months elsewhere in the body (""significant"" meaning 5 or more days in any month or any pain during the past month), e.g., low back pain, fibromyalgia, migraine headaches
5. Not meeting any of the most common pain-related TMD diagnoses as described in the DC/TMD criteria (myalgia, arthralgia, headache attributed to TMD) upon clinical exam following the DC/TMD protocol

Chronic painful TMD cases:

1. Primary TMD case criteria: Myalgia (masticatory muscle pain) based on clinical exam following the DC/TMD protocol
2. Concurrent arthralgia (TMJ pain) and/or headache attributed to TMD allowed
3. Myofascial pain must meet the following criteria:

   1. Onset >3 months, occurring >15 days/month on average for >3 months
   2. Minimum of 10 jaw pain episodes since onset, each lasting at least 30 minutes and no less than 2 hours within the day, OR unremitting."

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Traumatic facial injury or surgery on the face/jaw, arms, or hands
2. Presence of pain related to dental and periodontal pathology
3. Pregnant
4. Has any of the following medical conditions by self-report:

   1. Renal failure or dialysis
   2. Heart disease (examples: uncontrolled arrhythmia or hypertension, cardiomyopathy) or heart failure
   3. Non-allergic bronchospasm (chronic obstructive pulmonary disease and emphysema)
   4. Diabetes (type I or II) that is not controlled with medication or diet
   5. Hyperthyroidism
   6. Uncontrolled seizures
5. Used any injection therapy (e.g., tender or trigger point injections, steroid injections), acupuncture, biofeedback, or TENS for managing facial/jaw pain within 2 weeks before the screening assessment.
6. If undergoing botulinum toxin injections in the head and neck area, must be 3 months since the last set of injections, and refrain from this treatment until study participation has ended
7. History of major depression or other major psychiatric disorder requiring inpatient hospitalization within the last 6 months before the screening assessment
8. History of treatment for drug or alcohol abuse within the last 12 months
9. Current pain medication use (e.g., opioids, ibuprofen, acetaminophen) that cannot be stopped <24 hours before each study visit
10. Other conditions/diseases associated with altered pain perception: neurological or development disorders (dementia, autism spectrum disorder), neoplasm, multiple sclerosis, trigeminal neuralgia
11. Adults lacking the capacity to provide informed consent for themselves
12. Unable to understand instructions for sensory testing in English.
13. Thermal threshold for Pain-50 (pre-determined at the beginning of visit 1) is outside the temperature range of 40ºC to 49ºC
14. Inability to complete at least four daily ratings between the Informed consent, Pre-visit 1 procedures, and in-person visit 1
15. Lack of access to electronic devices with internet connection during the study participation
16. Anything that would place the individual at increased risk or preclude the individual's full compliance with study procedures or completion of the study. "

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: "1- Chronic Temporomandibular disorder (TMD) pain group 2- Age- and sex-matched pain-free controls"
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Conditioned pain modulation (CPM) effect | 3.5 hours single in-person visit
  The CPM effect is manifested as a reduction of pain intensity evoked by a test stimulus (Ts) presented concurrently or right after a painful conditioning stimulus (Cs) applied to a distant body site.
The relationship between daily pain intensity fluctuation and endogenous pain modulation (EPM) efficiency | 14 days: 7 days before and 7 days after the in-person visit
  The daily presentation of chronic TMD pain is variable, especially in those presenting with pain that affects their daily activities. This variability could be partially attributed to the varying efficiency of EPM in this patient population.

CONTACTS AND LOCATIONS:
Overall Officials: Estephan Moana-Filho, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States